CLINICAL TRIAL: NCT02669069
Title: Treatment Evaluation of Neuromodulation for Tinnitus (TENT-A)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromod Devices Ltd. (Industry)
Collaborators: University Hospital Regensburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neuromoddevices; TENT-A1 (Stage A1) (Other: Neuromod Devices Ltd.)
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Tinnitus
Keywords: Bi-modal neuromodulation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PS1 (Active Comparator)
  Interventions: Device: PS1
- PS2 (Active Comparator)
  Interventions: Device: PS2
- PS3 (Active Comparator)
  Interventions: Device: PS3

INTERVENTIONS:
Device: PS1 — Participants in this arm shall be given an audio stimulus which comprises of a sequence of tones, mixed with a broadband noise that is spectrally modified to compensate for any hearing loss. Electrical pulses in the somatosensory stimulation are synchronous with the tones.
  Arms: PS1
Device: PS2 — Participants in this arm shall be given an audio stimulus which comprises of a sequence of tones, mixed with a broadband noise that is spectrally modified to compensate for any hearing loss. Electrical pulses in the somatosensory stimulation are uncorrelated and asynchronous with the tones.
  Arms: PS2
Device: PS3 — Participants in this arm shall be given an audio stimulus which comprises of a sequence of single-frequency tones mixed with a broadband noise with the frequency characteristics of both chosen outside the region of any hearing loss. Electrical pulses in the somatosensory stimulation are uncorrelated and asynchronous with the tones.
  Arms: PS3

SUMMARY:
This is a three arm, patient subtyping and parameter optimisation study for a neuromodulation treatment for tinnitus.

DETAILED DESCRIPTION:
Participants with chronic tinnitus will be provided with a CE marked neuromodulation device. Devices will be programmed with one of 3 stimulation parameter settings. After 12 weeks of use, differences in tinnitus severity scores will be compared between the 3 arms and within the arms for patient subtype analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* The ability to read and understand English/German
* Willing and able to provide informed consent
* Willing to commit to the full duration of the study
* Have been experiencing tinnitus 3 months to 5 years
* Experiencing subjective tinnitus
* Baseline Tinnitus Handicap Inventory (THI) score of 28 to 76 points
* Baseline Minimum Masking Level (MML) of 20 to 80 dBHL
* Maximum AC pure-tone audiometry hearing loss of 80 dB HL at any test frequency in the range of 2 to 8 kHz or of 40 dB HL in the range of 250 to 1000 Hz either unilaterally or bi-laterally

Exclusion Criteria:

* If participant has been diagnosed with objective tinnitus
* Commenced usage of hearing aid within the last 90 days
* Cases where pulsatility is the dominant feature of tinnitus
* Patients whose tinnitus cannot be masked during MML assessment
* Meniere's disease
* Significantly severe Loudness Discomfort Level (LDL), <30 dB SL
* Depression or neuro-psychological condition, previously diagnosed or identified from the State-Trait Anxiety Inventory (STAI) scores greater than 120
* Diagnosed with somatic tinnitus resulting from head or neck injury
* Temporomandibular Joint Disorder (TMJ)
* Current or previous involvement in medico-legal cases
* Pregnancy
* Oral piercings
* Neurological conditions that may lead to loss of consciousness (e.g. epilepsy) or is considered to be the dominant feature of the tinnitus, as assessed by audiologist or ENT consultant
* Severe cognitive impairment based on Mini Mental State Examination (MMSE), less than 20
* Pacemakers or other electro-active implanted devices
* Have used Neuromod Devices products in the past
* Participants currently prescribed drugs for a Central Nervous System pathology, i.e. epilepsy, Multiple Sclerosis (MS), Parkinson's, bi-polar disorder.
* The site Principal Investigator does not deem the candidate to be suitable for the study for other reasons not listed above
* Self-reporting episodes of Auditory hallucinations
* Abnormal Otoscopy as assessed by the Audiologist, including active Otitis Media, perforation and hearing loss that is identified as completely conductive
* Abnormal Tympanometry as assessed by the Audiologist

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Tinnitus Functional Index | Between baseline and 12 weeks
Tinnitus Handicap Inventory | Between baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mr. Brendan Conlon, Principal Investigator — St. James's Hospital, Ireland; Prof. Dr. med. Berthold Langguth, Principal Investigator — University of Regensburg
Locations (2):
- University Hospital Regensburg, Regensburg, Germany
- St. James's Wellness Trust Clinical Research Facility, Dublin, Ireland

REFERENCES:
- [Background] D'Arcy S, Hamilton C, Hughes S, Hall DA, Vanneste S, Langguth B, Conlon B. Bi-modal stimulation in the treatment of tinnitus: a study protocol for an exploratory trial to optimise stimulation parameters and patient subtyping. BMJ Open. 2017 Oct 25;7(10):e018465. doi: 10.1136/bmjopen-2017-018465. PMID 29074518
- [Result] Conlon B, Langguth B, Hamilton C, Hughes S, Meade E, Connor CO, Schecklmann M, Hall DA, Vanneste S, Leong SL, Subramaniam T, D'Arcy S, Lim HH. Bimodal neuromodulation combining sound and tongue stimulation reduces tinnitus symptoms in a large randomized clinical study. Sci Transl Med. 2020 Oct 7;12(564):eabb2830. doi: 10.1126/scitranslmed.abb2830. PMID 33028707